CLINICAL TRIAL: NCT04230395
Title: Hybrid Trial for Alcohol Reduction Among People With TB and HIV in India (HATHI)
Brief Title: Alcohol Reduction Among People With TB and HIV in India
Acronym: HATHI
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IRB00235134; R01AA027974 (NIH)
Record Dates: First submitted 2020-01-14; First posted 2020-01-18 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Tuberculosis; HIV
Keywords: Alcohol Use; HIV; Tuberculosis
MeSH Terms: conditions — Tuberculosis; Alcohol Drinking

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HATHI (Experimental): The HATHI intervention is an up to 4-session alcohol reduction intervention that uses a combination of Motivational Enhancement Therapy and Cognitive Behavioral Therapy. The intervention will also include 3 booster sessions.
  Interventions: Behavioral: HATHI Intervention
- Usual Care (Other): Provider advice to reduce alcohol use per recommended standard of clinical care, and referral to treatment as indicated
  Interventions: Other: Usual Care

INTERVENTIONS:
Behavioral: HATHI Intervention — 4-session combination Motivational Enhancement Therapy and Cognitive Behavioral Therapy alcohol reduction intervention. The intervention will also include 3 booster sessions.
  Arms: HATHI
Other: Usual Care — Provider advice to reduce alcohol use per recommended standard of clinical care, and referral to treatment as indicated
  Arms: Usual Care

SUMMARY:
The highest incidence of tuberculosis disease (TB) in the world is in India, accounting for 27% of all new cases globally, with approximately 86,000 among persons with HIV (PWH). Unhealthy alcohol use can worsen the health of people who have Tuberculosis (TB), HIV and people who have both TB and HIV. Behavioral interventions that 1) target alcohol use and 2) are integrated into TB and TB/HIV and HIV care may lead to better outcomes. The goal of this study is to test if a behavioral alcohol reduction intervention integrated into TB, TB/HIV and HIV treatment can reduce alcohol use and improve TB and HIV health outcomes among people with unhealthy alcohol use. The aims of the HATHI study are: Aim 1: To test if a 4 session behavioral alcohol reduction intervention, called HATHI, integrated into TB and TB/HIV and HIV Care can decrease unhealthy alcohol use among persons with TB and TB/HIV coinfection and HIV. Aim 2: To test if the HATHI intervention, integrated into TB and TB/HIV and HIV care can improve TB and HIV clinical outcomes; Aim 3: To evaluate barriers and facilitators to integrating HATHI intervention into TB and TB/HIV and HIV care, and to determine the incremental costs of delivering HATHI intervention in TB and HIV clinical settings. Investigators hypothesize that HATHI intervention will reduce alcohol use among persons with TB and TB with HIV and HIV, and that its delivery in the TB and HIV setting will be acceptable to patients and providers and feasible.

DETAILED DESCRIPTION:
In 2017, over 10 million people worldwide developed tuberculosis disease (TB), with 9% of cases among people with HIV (PWH). In that same year, there were 1.6 million deaths from TB, with 300,000 among PWH. The highest incidence of TB is in India, accounting for 27% of all new cases globally, with approximately 86,000 among PWH. Unhealthy alcohol use triples the risk of TB in the general population, increasing susceptibility to primary infection and reactivation. Among PWH, unhealthy alcohol use is associated with decreased use of and adherence to antiretroviral therapy (ART), lower viral suppression and increased mortality. Treatment for TB presents a unique opportunity to address unhealthy alcohol use among people with TB and TB/HIV coinfection and HIV given the frequent contact participants have with healthcare providers and the deleterious effects of unhealthy use on both HIV and TB clinical outcomes. Although combined cognitive behavioral therapy (CBT) and motivational enhancement therapy (MET) can be effective in reducing alcohol use, access to and implementation of such interventions is limited in high-need, under-resourced low and middle income (LMIC) settings. Even in settings where formal treatment is available, alcohol-related stigma and cost of treatment may prevent individuals from seeking care. Integrating treatment for unhealthy alcohol use into TB and TB/HIV and HIV care may overcome barriers to alcohol treatment for such individuals at risk for poor health outcomes. HATHI (Hybrid trial for Alcohol reduction among people with TB, TB/HIV and HIV in India), is a 2-arm hybrid type 1 effectiveness-implementation randomized controlled trial (RCT) examining the effectiveness of a four-session combined CBT/MET alcohol reduction intervention (HATHI), followed by three intervention boosters, integrated into TB and TB/HIV and TB care, compared with usual care (provider advice, referral to treatment as needed). There will be 3 phases. In Phase 1) investigators will tailor the intervention based on results from a) focus groups (FG) with patients with TB and HIV, medical and clinical staff, and the intervention counselors (IC) and b) individual intervention testing with a subgroup of patients with TB and HIV. In Phase 2) investigators will conduct an RCT in which participants will be randomized to HATHI intervention or to usual care. Investigators will stratify persons with TB/HIV coinfection by HIV status to ensure balance of HIV between the groups. Effectiveness outcomes measured at 3, 6 and 12 months will include 1) phosphatidyl ethanol (PEth), an alcohol biomarker (primary), and self reported alcohol use (secondary) 2) TB and HIV clinical outcomes. In Phase 3, evaluating trial participants, counselors, clinical and organizational staff, investigators will use the RE-AIM implementation framework using mixed methods to assess barriers and facilitators to alcohol treatment integration in TB and HIV clinical settings and to assess the incremental costs of this intervention strategy.

Setting: All phases of the study will take place at two sites in India: the Byramjee Jeejeebhoy Government Medical College (BJGMC) and Dr. DY Patil Medical College, Pune (DYPMC).

Objectives/Aims:

Aim 1: In a randomized controlled trial (RCT), to examine the effectiveness of CBT/MET integrated into TB, TB/HIV and HIV care compared to usual care on alcohol use.

Aim 2: In a RCT, to examine the effectiveness of CBT/MET integrated into TB, TB/HIV and HIV care compared to usual care on TB and HIV treatment outcomes.

Aim 3: Guided by the RE-AIM implementation framework, and using mixed methods, to 3a) evaluate patient, provider and organizational barriers and facilitators to integrated alcohol treatment in TB and HIV settings, and 3b) measure incremental costs from health system and societal perspectives.

Prior to RCT implementation investigators will tailor HATHI and make final modifications to the HATHI manual. HATHI will be enhanced with content specific to Pune such as local alcohol containing beverages and local or state drinking norms and alcohol impacts on TB and HIV progression and clinical outcomes. Investigators will modify the manual and test in focus groups.

Phase 2-Clinical Trial. This phase involves collection of routinely used research assessments for individuals with TB and TB/HIV and HIV at baseline, 3, 6, and 12 months and the launch of the RCT. The study will include adults individuals with 1) newly diagnosed TB (with or without HIV), unhealthy alcohol use, initiating TB medication treatment and 2) persons with HIV and unhealthy alcohol use. Individuals will be recruited through both provider and self-referral. Up to half of the sample will have both TB and HIV. Eligible individuals will undergo baseline assessment which includes a medical history, clinical exam, questionnaires, and a blood spot for the alcohol biomarker PEth.

Assignments of Participants to the Study Intervention: Eligible participants will be randomized in a 1:1 ratio upon completion of the baseline evaluation. The study biostatistician, independent of the trial will generate the randomization sequence in permuted blocks and randomization of persons with TB will be stratified by the presence of HIV infection. A sealed envelope with study assignment will be used to conceal the study group assignment.

Study Conditions:

Control: Individuals in the control arm will receive standard of care TB and HIV treatment and usual care from participants' provider, which includes advice to reduce alcohol use and referral to alcohol treatment services at participants' provider's discretion.

Intervention: HATHI is an up to 4-session manualized alcohol reduction treatment based on Cognitive Behavioral and Motivational Enhancement Therapy. Each session lasts up to 45 minutes. The 4 HATHI sessions will be delivered by a counselor during an 8 week period, closely aligned to regular TB treatment follow up visits. After the 4 intervention sessions, individuals will receive 3 scripted booster sessions, one month apart, corresponding to participants' follow up visits.

Research Data Ascertainment: Assessments will occur at baseline (prior to randomization), 3 months (end of 4 session intervention), 6, and 12 months post-baseline. Data collection will include self-report questionnaires staff interviews, and biomarker and specimens and will encompass demographics, a clinical assessment, measurement of alcohol use, its severity and consequences; HIV measures including viral load, medication adherence and HIV retention in care; TB measures, including TB clearance, TB treatment default, TB medication adherence and TB retention in care. Other measures span mental health, tobacco and other substance use, quality of life, diabetes mellitus, motivation to change and self-efficacy.

Investigators' primary alcohol endpoint will occur at 6 months after baseline, with investigators' secondary endpoint at 12 months. Sample size calculations are based on data from behavioral alcohol reduction interventions in low and middle income countries.

Investigators' trial will enroll a total of 450 participants with TB or TB/HIV or HIV; The study will be conducted at two sites and 2 counselors at each site will administer the intervention. Power calculations assume a 10% loss to follow-up, and intra-class correlation coefficient of 0.04 (based on Counseling on Alcohol Problems (CAP)/PREMIUM RCT) to account for 2 counselors per site, 2 sites). Analyses will also account for variation by counselor and by site.

Phase 3: The Reach, Effectiveness, Adoption, Implementation, and Maintenance (RE-AIM) implementation framework will be used to collect quantitative and qualitative assessments from 3 levels of stakeholders (Numbers approximate, pending thematic saturation). Investigators will evaluate barriers and facilitators to intervention reach, effectiveness, adoption, implementation and maintenance, focusing in implementation outcomes of feasibility, acceptability, appropriateness, fidelity and sustainability. Investigators will also calculate the incremental costs of the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Active TB defined as either a) microbiologically confirmed TB (sputum AFB smear positive by microscopy or +GeneXpert at entry) or b) clinical TB that is subsequently confirmed by Acid-Fast Bacilli (AFB) culture; with or without concurrent HIV infection)
* HIV infection
* initiating TB therapy;
* age ≥ 18 years of age;
* AUDIT Score ≥ 8 in men /≥ 6 in women.

Exclusion Criteria:

* already in treatment for unhealthy alcohol use;
* unable to participate in intervention sessions either due to severity of medical illness, cognitive dysfunction or active psychosis;
* pregnant (will refer directly to alcohol treatment)
* household member of current study participant
* Patients reported to have Drug Resistant TB, Multidrug-Resistant Tuberculosis (MDR-TB) and Extrapulmonary tuberculosis (EPTB) if they are in only TB cohort.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 450 (Estimated)
Dates: Start 2022-09-22 (Actual); Primary Completion 2026-02-15 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
PEth | 6 months
  PEth biomarker will be used as a liner variable and log transformed if data are skewed

SECONDARY OUTCOMES:
Change in Alcohol Use as assessed by change in Drinking days | 3 months and 12 months
  Change in Self reported number of drinking days on the 30-day Time Line Follow Back Interview (TLFB)
Change in Alcohol Use as assessed by change in heavy Drinking days | 3 months and 12 months
  Change in Self reported heavy drinking days on the 30-day Time Line Follow Back Interview (TLFB)
Change in Alcohol Use as assessed by change in standard drinks per drinking days | 3 months and 12 months
  Change in Self reported standard drinks per drinking day on the 30-day Time Line Follow Back Interview
TB treatment failure, TB treatment default, or all-cause mortality | 12 months
  Composite outcome: TB treatment failure, TB treatment default, or all-cause mortality (defined as a binary outcome i.e. 0=none of these outcomes and 1= one or more of these outcomes)
HIV-RNA Non-Suppression | 6 months
  This will be assessed as HIV-RNA >200 copies
HIV-RNA Non-Suppression | 12 months
  This will be assessed as HIV-RNA >200 copies
Alcohol Use: Drinking days | 6 months
  Self reported number of drinking days on the 30-day Time Line Follow Back Interview (TLFB)
Alcohol Use: Heavy drinking days | 6 months
  Self reported heavy drinking days on the 30-day Time Line Follow Back Interview (TLFB)
Alcohol Use: Standard drinks per drinking day | 6 months
  Self reported standard drinks per drinking day the 30-day Time Line Follow Back Interview (TLFB)

OTHER OUTCOMES:
Change in Phosphatidyl Ethanol | 3, 6, 12 months
  We will assess change in blood levels of Phosphatidyl Ethanol as an Alcohol Biomarker

CONTACTS AND LOCATIONS:
Overall Officials: Amita Gupta, MD, Principal Investigator — Johns Hopkins University
Locations (2):
- India (2):
  - BJ Government Medical College and Sassoon General Hospital, Pune, Maharashtra
  - Dr. D. Y. Patil Medical College, Pune, Maharashtra

IPD SHARING:
Plan to Share IPD: Yes
Per NOT-AA-19-020, we will share/upload data to the NIAAA Data Archive (NIAAADA).